CLINICAL TRIAL: NCT04126473
Title: A Phase 2 Open Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Dose Levels of Subcutaneously Administered ELX-02 in Patients With Cystic Fibrosis With at Least One G542X Allele
Brief Title: A Phase 2 Study to Evaluate the Safety, Tolerability, PK and PD in Cystic Fibrosis Patients With at Least 1 G542X Allele
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eloxx Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EL-004
Record Dates: First submitted 2019-08-16; First posted 2019-10-15 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
Keywords: aminoglycoside; Nonsense Mutation; Translational read through
MeSH Terms: conditions — Cystic Fibrosis | interventions — ELX-02; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ELX-02 (Experimental): Eukaryotic ribosomal selective glycoside (ERSG)
  Interventions: Drug: ELX-02; Drug: Ivacaftor

INTERVENTIONS:
Drug: ELX-02 — ELX-02 is a small molecule, new chemical entity being developed for the treatment of genetic diseases caused by nonsense mutations. ELX-02 is a eukaryotic ribosomal selective glycoside (ERSG).
Drug: Ivacaftor — CFTR potentiator

SUMMARY:
This is a Phase 2 open label study to evaluate the safety, tolerability, PK, and PD of multiple dose levels of SC administered ELX-02 with and without ivacaftor in patients with CF with at least one G542X allele or phenotypically similar nonsense allele.

Up to 16 patients will be enrolled in the trial; up 4 patients will be homozygotes to G542X, and the remaining patients will be compound heterozygotes with G542X or phenotypically similar nonsense mutation and any Class 1 or Class 2 mutation.

Each patient will receive 5 escalating doses as follows:

* 0.3 mg/kg per day SC
* 0.75 mg/kg per day SC
* 1.5 mg/kg per day SC
* An individualized dose, as high as 3.0 mg/kg per day SC, based upon the patients observed safety and tolerability, PK at previous doses and the results of laboratory tests
* ELX-02 1.5 mg/kg per day SC plus 150 mg ivacaftor every 12 bid

ELIGIBILITY:
Patients must meet the following criteria to participate in this study:

1. Males and females age 18 years and above in Germany and Israel; in countries where permitted, males and females age 16 years and above
2. A confirmed diagnosis of nmCF with a documented G542X or phenotypically similar nonsense mutation, homozygote, or compound heterozygote with one of the specified mutations. For heterozygotes, one mutation has to be G542X or phenotypically similar nonsense mutation, and the second mutation could be and Class 1 or Class 2 mutation. Patients with one G542X or phenotypically similar nonsense allele and a second allele that is not in the above list may be potentially allowed but only after discussion on a case by case basis with and written approval from the Sponsor.
3. Documented SCC ≥ 60 mEq/L
4. FEV1 ≥ 40% predicted normal for age, gender and height at Screening (Knudson Equation)
5. Body Mass Index (BMI) of 19.0 to 30.0 kg/m2 (inclusive).

Patients with any of the following characteristics/conditions will not be included in the study:

1. Participation in clinical study including administration of any investigational drug or device in the last 30 days or 5 half-lives (whichever is longer) prior to investigational product dosing in the current study
2. History of any organ transplantation
3. Major surgery within 180 days (6 months) of Screening
4. Patients without documented prior aminoglycoside exposure who have a mitochondrial mutation that has been shown to increase sensitivity to aminoglycosides
5. Known allergy to any aminoglycoside
6. Patients with any abnormality at ENT screening, that indicates the presence of a vestibular toxicity associated with prior exposure to aminoglycosides.
7. Dizziness Handicap Inventory (DHI)-H score at screening >16
8. Patients receiving CFTR modulators within 2 months of study treatment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
AEs associated with different dose levels of ELX-02 | From the time of first dosing through the follow-up visit, an average of approximately 9 weeks
Area under the plasma concentration curve from time zero to 24 hours (AUC0-24) | Day 1 of treatment periods 1, 2, 3, and 4
  Full PK profile 8 blood samples up to 24 hours
Maximum observed plasma concentration (Cmax) on Day 1 | Day 1 of treatment periods 1, 2, 3, and 4
  Full PK profile 8 blood samples over 24 hours
Peak observed plasma concentration (Cpeak) over time | Days 1, 2 and 7 of treatment periods 1-3, Days 1, 2, 7, and 14 of treatment period 4, sparse sampling, blood sampling at 30 min and 1 hour post-dose
Trough observed plasma concentrations (Cpredose) over time | Days 1, 2 and 7 of treatment periods 1-3, Days 1, 2, 7 and 14 of treatment period 4, sparse blood sampling at pre-dose

SECONDARY OUTCOMES:
Changes from baseline in sweat chloride concentration | From baseline to Day 7 of treatment periods 1-3, and Days 7 and 14 of treatment period 4
Changes from baseline in percent predicted forced expiratory volume (ppFEV1) | From baseline to Day 7 of treatment periods 1-3, and Days 7 and 14 of treatment period 4
Changes from baseline in percent predicted forced vital capacity (ppFVC) | From baseline to Day 7 of treatment periods 1-3, and Days 7 and 14 of treatment period 4
Changes from baseline in percent predicted forced expiratory flow at 25-75% (ppFEF25-75) | From baseline to Day 7 of treatment periods 1-3, and Days 7 and 14 of treatment period 4

CONTACTS AND LOCATIONS:
Locations (9):
- Australia (3):
  - The Royal Prince Alfred Hospital, Camperdown, New South Whales
  - The Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- Germany (2):
  - Universitätsmedizin Essen Ruhrlandklinik, Essen, North Rhine-Westphalia
  - Universitätsklinikum Frankfurt, Frankfurt
- Israel (4):
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Schneider Children's Medical Center, Petach Tikvah
  - Safra Children's Hospital - Chaim Sheba Medical Center, Ramat Gan

REFERENCES:
- See also: Eloxx Pharmaceuticals Website — http://www.eloxxpharma.com